CLINICAL TRIAL: NCT03222648
Title: Investigating the Effects of a Structured Responsive Exercise Training Programme in Idiopathic Pulmonary Fibrosis - a Pilot Study
Brief Title: Structured Exercise Training Programme in Idiopathic Pulmonary Fibrosis
Acronym: Rehab-IPF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Timothy Wallis, Doctor, University Hospital Southampton NHS Foundation Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHM MED1441
Record Dates: First submitted 2017-06-23; First posted 2017-07-19 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Breathlessness; Quality of Life; Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; Exercise training; Health related quality of life; Biomarkers
MeSH Terms: conditions — Dyspnea; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: single cohort pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Responsive Exercise Training (Experimental): 8 week twice weekly supervised structured responsive static-cycle based exercise training. Training protocol used the same as Loughney et al. 2016
  Interventions: Other: Structured Responsive Exercise Training
- Standard of Care Arm (Active Comparator): Completion of outcome measures only
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Structured Responsive Exercise Training — Twice weekly, 8 week structured responsive exercise training programme. Protocol used the same as that used in previous EMPOWER Trial (Loughney et al. 2016)
  Arms: Structured Responsive Exercise Training
Other: Usual Care — Continuation of usual care
  Arms: Standard of Care Arm

SUMMARY:
In this single centre non-randomised pilot cohort study we wish to quantify the effect of a twice weekly, 8 week, structured responsive exercise training programme on exercise tolerance, symptoms and health related quality of life in patients with Idiopathic Pulmonary Fibrosis (IPF). We also wish to assess the effect of exercise training on fibrotic processes causing IPF through measurement of blood biomarkers of disease activity.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is a progressive fibrotic lung disease characterised by progressive exercise intolerance and breathlessness. In 2012 there were 32 500 people living in the United Kingdom (UK) with IPF. Average life expectancy from time of diagnosis is 2-3 years (Ley et al. 2011). Despite recent advances in drug therapy, therapeutic options are limited and no medication has been found to halt progression of the disease. Pulmonary Rehabilitation (PR) is a structured exercise and education intervention that is well established as a core treatment intervention for patients with Chronic Obstructive Pulmonary Disease (COPD). Current limited evidence shows that PR is safe in patients with IPF and can lead to short-term improvements in exercise tolerance, symptoms and quality of life (Dowman et al. 2014). However the optimal exercise protocol, the longer-term benefits and which group or patients (those with milder or more severe disease) benefit most is unclear. Further it is unknown what mechanisms underlie any improvement and whether exercise training influences the fibrotic process causing IPF.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18-85 years with a confirmed diagnosis of fibrotic interstitial lung disease (fILD) including; Usual Interstitial Pneumonia, fibrotic Nonspecific interstitial pneumonia (NSIP), Chronic hypersensitivity pneumonitis (chronic HP) and unclassifiable interstitial lung disease (unclassified ILD). Medical Research Council (MRC) breathlessness scale grade 1-3. Clinically stable for 3 months as judged by investigator

Exclusion Criteria:

* Forced Expiratory Volume in 1 second (FEV1) to Forced Vital Capacity (FVC) FEV1/FVC ratio <0.7
* Patients with severe heart failure New York Heart Association (NYHA) grade III or IV or left ventricular systolic function <45%
* Current use of ambulatory or long term oxygen therapy
* Resting oxygen saturations <85% on air
* The presence of infection or exacerbation requiring hospitalization, within 3 months prior to recruitment
* Commencement on anti-fibrotic therapy (Pirfenidone® or Nintedanib®) within 3 months prior to recruitment to the study
* Patients taking oral corticosteroids: unless the dose is less than 15 mg of prednisolone or equivalent, and the dose has been stable for 8 weeks at the time of booking
* Neoplastic disease undergoing treatment or active follow-up
* Current or previous history of sarcoidosis or collagen vascular disease
* Any condition which would prevent completion of cycle-ergometer testing, Pulmonary Function Tests (PFTs) or 6 minute walk test (6-MWT) as judged by the investigator.
* Participation in a Pulmonary Rehabilitation (PR) program in the last 6 months
* Any condition excluding Cardiopulmonary Exercise Testing (CPET) based on the absolute contraindication as the American College of Chest Physicians (ACCP)/ American Thoracic Society (ATS) guidelines 2003 listed here: History of exercise induced syncope, Uncontrolled arrhythmia causing symptoms or hemodynamic compromise, Syncope, Acute endocarditis, Acute myocarditis or pericarditis, Symptomatic severe aortic stenosis, Uncontrolled heart failure, History of acute venous thrombo-embolism, Suspected dissecting aneurysm, uncontrolled asthma, Pulmonary oedema, Mental impairment leading in ability to cooperate, Room air desaturation to <85% unless supplemental O2 is provided for exercise, Acute non-cardiopulmonary disorder that may affect exercise performance/ aggravated by exercise
* Positive Pregnancy test in females of childbearing age.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in endurance time on fixed load cycle | 8 weeks
  validated fixed load static cycling test at 75% peak oxygen consumption (VO2 peak) derived from derived from cardiopulmonary exercise testing (CPET) (seconds)

SECONDARY OUTCOMES:
Change from baseline in St. George's Respiratory Questionnaire -IPF (SGRQ-I) | 8 weeks
  Validated health and quality of life questionnaire for patients with IPF
Change from baseline in Medical Research Council (MRC) Breathlessness Scale | 8 weeks
  Validated breathlessness questionnaire for respiratory patients
Change from baseline in Revised Borg Breathlessness Score | 8 weeks
  Validated breathlessness score for respiratory patients
Change from baseline in 6 - Minute Walk Test Distance | 8 weeks
  Validated exercise capacity assessment for respiratory patients (meters)
Change from baseline Cardiopulmonary Exercise Test variables | 8 weeks
  A validated tool for access multiple parameters of exercise capacity measures including but not limited to; peak Oxygen consumption ml/kg/minute (VO2 peak), anaerobic threshold ml/kg/minute (AT) , volume of oxygen work rate relationship ml/watt (VO2/Work Rate)
Change from baseline in Fat Mass Index (FMI) | 8 weeks
  measured by Bioelectrical Impedance Analysis a validated tool to access multiple parameters of body composition.
Change from baseline in Phase Angle measured by | 8 weeks
  measured by Bioelectrical Impedance Analysis a validated tool to access multiple parameters of body composition.
Change from baseline in Fat Free Mass Index (FFMI) | 8 weeks
  measured by Bioelectrical Impedance Analysis a validated tool to access multiple parameters of body composition.
Change from baseline in Skeletal Muscle Mass (kg) | 8 weeks
  measured by Bioelectrical Impedance Analysis a validated tool to access multiple parameters of body composition.
Change from baseline in Body Mass Index (kg/m2) | 8 weeks
  weight (kg)/height (m)2.
Change from baseline in Council of Nutrition Appetite Questionnaire (CNAQ) | 8 weeks
  A validated nutritional assessment tool. CNAQ Total Score 8-40 (40 better outcome)
Change from baseline in Simplified nutritional appetite questionnaire (SNAQ) questionnaire | 8 weeks
  A validated nutritional assessment tool. SNAQ 5-20 (20 better outcome)
Change from baseline in EQ-5D-5L | 8 Weeks
  A validated global health related quality of life PROM. Total Score, Subsections (Mobility, Self-Care, Usual Activity, Pain/Discomfort, Anxiety/Depression. Visual Analogue Scale (0-100)

OTHER OUTCOMES:
Change from baseline in Blood biomarkers of disease activity in Idiopathic Pulmonary Fibrosis | 8 weeks
  Plasma/Serum biomarkers including but not limited to Surfactant protein D, Periostin, Matrix Metalloproteinase-7 (MMP-7) and collagen neoepitopes.
Change from baseline in Blood markers of oxidative stress | 8 weeks
  Plasma markers of oxidative stress including but not limited to 15-F2t-isoprostanes
Change from baseline in serum albumin | 8 weeks
  Blood markers of systemic inflammation
Change from baseline in serum C-Reactive Protein | 8 weeks
  Blood markers of systemic inflammation
Change from baseline in serum Interleukin-8 | 8 weeks
  Blood markers of systemic inflammation
Change from baseline in total white blood cell count | 8 weeks
  Blood markers of systemic inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Tim JM Wallis, MA BM MRCP, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loughney L, West MA, Kemp GJ, Rossiter HB, Burke SM, Cox T, Barben CP, Mythen MG, Calverley P, Palmer DH, Grocott MP, Jack S. The effects of neoadjuvant chemoradiotherapy and an in-hospital exercise training programme on physical fitness and quality of life in locally advanced rectal cancer patients (The EMPOWER Trial): study protocol for a randomised controlled trial. Trials. 2016 Jan 13;17:24. doi: 10.1186/s13063-015-1149-4. PMID 26762365
- [Background] Ley B, Collard HR, King TE Jr. Clinical course and prediction of survival in idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2011 Feb 15;183(4):431-40. doi: 10.1164/rccm.201006-0894CI. Epub 2010 Oct 8. PMID 20935110
- [Background] Dowman L, Hill CJ, Holland AE. Pulmonary rehabilitation for interstitial lung disease. Cochrane Database Syst Rev. 2014 Oct 6;(10):CD006322. doi: 10.1002/14651858.CD006322.pub3. PMID 25284270